CLINICAL TRIAL: NCT04954872
Title: Comparing Strategies for Competency-based Training in Problem Management Plus to Improve Non-specialist Competencies for Responding to Psychological Distress: a Randomized Controlled Trial
Brief Title: Competency-based Training in Problem Management Plus: a Randomized Controlled Trial
Acronym: EQUIP-PM+
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: George Washington University (Other)
Collaborators: Transcultural Psychosocial Organization Nepal (Other)
Responsible Party: Principal Investigator, Brandon A Kohrt, MD, PhD, Professor, George Washington University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: NCR191797-v2
Record Dates: First submitted 2021-06-29; First posted 2021-07-08 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Depression
Keywords: Training; Competency; Psychological treatment
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: Persons without mental health professional experience will be randomized to either training as usual to develop Problem Management Plus competencies or they will be randomized to Problem Management Plus training that uses Equip principles of competency-based training.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: The persons without mental health professional training who are randomized to either training as usual or Equip-based training will not be informed about how the two training arms differ. Outcome assessors will not be told if the trainees are in training as usual or Equip-based training.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training as usual (Active Comparator): Standard Problem Management Plus training.
  Interventions: Behavioral: Standard Problem Management Plus training (training as usual)
- Equip-based training (Experimental): Training that uses the Equip platform to assess competencies and incorporate this information into trainers and supervisors activities.
  Interventions: Behavioral: Equip-based Problem Management Plus training

INTERVENTIONS:
Behavioral: Standard Problem Management Plus training (training as usual) — 10-day training on Problem Management Plus.
  Arms: Training as usual
Behavioral: Equip-based Problem Management Plus training — Training and supervision for Problem Management Plus in which the trainers and supervisors use the EQUIP platform for competency assessment and feedback.
  Arms: Equip-based training

SUMMARY:
The proposed study in Nepal will evaluate if non-specialists participating in Equip-based Problem Management Plus training show greater competencies compared to non-specialists participating in standard Problem Management Plus training. The proposed study is a randomized controlled trial with mixed-methods components evaluating both quantitative outcomes and qualitative outcomes among non-specialists participating in the training and their trainers.

DETAILED DESCRIPTION:
There is increasing recognition of the high burden of psychological distress among populations around the world. Increasingly, non-specialists (persons who do not have expertise in formal mental health training) are being used to deliver psychological services. There is a long history of successful implementation of psychological services by non-specialists in Nepal. Recently, a cluster randomized controlled trial of Problem Management Plus showed modest benefit over enhanced care as usual in southeastern Nepal. A recent initiative by the World Health Organization is being rolled out to improve the competencies of non-specialists participating in Problem Management Plus and similar trainings. This initiative is Ensuring Quality in Psychological Services (Equip). The proposed study in Nepal will evaluate if non-specialists participating in Equip-based Problem Management Plus training show greater competencies compared to non-specialists participating in standard Problem Management Plus training. The proposed study is a randomized controlled trial with mixed-methods components evaluating both quantitative outcomes and qualitative outcomes among non-specialists participating in the training and their trainers.

ELIGIBILITY:
Inclusion Criteria:

* No prior mental health professional training
* Literate in Nepali

Exclusion Criteria:

* Any prior mental health professional training

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Enhancing Assessment of Common Therapeutic Factors (unabbreviated title: Enhancing Assessment of Common Therapeutic Factors) | Immediately after Problem Management Plus training (10-days post-baseline)
  15-item tool with 4 response levels, range is 15 to 60, with higher scores equating to more competency

SECONDARY OUTCOMES:
Enhancing Assessment of Common Therapeutic Factors (unabbreviated title: Enhancing Assessment of Common Therapeutic Factors) | After Problem Management Plus supervision (approximately 45-days post-baseline)
  15-item tool with 4 response levels, range is 15 to 60, with higher scores equating to more competency
Problem Management Plus Competency Assessment (unabbreviated title: Problem Management Plus Competency Assessment) | Immediately after Problem Management Plus training (10-days post-baseline)
  12-item tool with 4 response levels, range is 12 to 48, with higher scores equating to more competency
Problem Management Plus Competency Assessment (unabbreviated title: Problem Management Plus Competency Assessment) | After Problem Management Plus supervision (approximately 45-days post-baseline)
  12-item tool with 4 response levels, range is 12 to 48, with higher scores equating to more competency
Group Facilitation Competency Assessment (unabbreviated title: Group Facilitation Competency Assessment) | Immediately after Problem Management Plus training (10-days post-baseline)
  8-item tool with 4 response levels, range is 8 to 32, with higher scores equating to more competency
Group Facilitation Competency Assessment (unabbreviated title: Group Facilitation Competency Assessment) | After Problem Management Plus supervision (approximately 45-days post-baseline)
  8-item tool with 4 response levels, range is 8 to 32, with higher scores equating to more competency

CONTACTS AND LOCATIONS:
Overall Officials: Brandon A Kohrt, MD, PhD, Principal Investigator — George Washington University
Locations (1):
- Transcultural Psychosocial Organization Nepal, Kathmandu, Nepal

IPD SHARING:
Plan to Share IPD: Yes
Researchers can contact the principal investigator for access to data.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After publication of primary results
Access Criteria: Submit a proposal for intended analysis to the principal investigator.